CLINICAL TRIAL: NCT02738320
Title: Patient Centered Quality Reporting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Dana Mukamel, Professor of Medicine, Public Health and Nursing, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: HS# 2012-9098
Record Dates: First submitted 2016-04-05; First posted 2016-04-14 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-04

CONDITIONS: Quality Report Cards

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Intervention (Experimental): Intervention patients will receive access to NHCPlus when discharge to a nursing home from the hospital is expected.
  Interventions: Other: NHCPlus
- Usual Care (No Intervention): Control patients will receive the usual care when discharge to a nursing home from the hospital is expected.

INTERVENTIONS:
Other: NHCPlus — A decision-aid tool that will interface with Nursing Home Compare and improve consumers' ability to assimilate and incorporate the information into their process of choosing a nursing home.
  Arms: Intervention

SUMMARY:
The purpose of this study is to develop a consumer friendly web-based interface between Nursing Home Compare (NHC) and an e-coaching/decision-aid tool (NHCPlus) and determine if use of NHCPlus facilitates and enhances access to and use of NHC.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have been admitted as an inpatient into the departments of Medicine or Surgery at the UC Irvine Medical Center, and whose discharge plan is to a nursing home.
* Family members of these patients, if they are involved in the choice of nursing home, were also recruited to the study, either as joint decision makers with the patients or as proxy decision makers for the patient.

Exclusion Criteria:

* Patients less than 50 years of age.
* Patients unable to use NHCPlus technology or participate in the nursing home choice decision (i.e. non-English speaking, severely visual or hearing impaired, dementia, or other debilitating illnesses) will be excluded unless they have a representative/proxy who will be involved in the decision to select the nursing home.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2014-03; Primary Completion 2015-09 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Use of Nursing Home Compare information | up to 9 days post discharge
  Patients (or their families) self report their knowledge and use of the information in Nursing Home Compare.
Quality Measures of chosen nursing home | up to 9 days post-discharge
  Quality measures obtained from the Nursing Home Compare web based report card
Distance between patient/family residence and the chosen nursing home. | up to 9 days post-discharge
  Driving distance between the patient zip code and the chosen nursing home zip code using Google maps.
Length of stay in hospital | between 1 and 68 days
  Number of days between admission date and discharge date

CONTACTS AND LOCATIONS:
Overall Officials: Dana Mukamel, PhD, Principal Investigator — University of California
Locations (1):
- University of California, Irvine, California, United States